CLINICAL TRIAL: NCT01585246
Title: Saw Palmetto Use During Radiation Therapy for Symptom Management Among Prostate Cancer Patients
Brief Title: Saw Palmetto: Symptom Management for Men During Radiation Therapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Michigan State University (Other)
Responsible Party: Principal Investigator, Gwen Wyatt, Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Application ID 213
Record Dates: First submitted 2012-04-23; First posted 2012-04-25 (Estimated); Results first posted 2017-07-14 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Radiation Therapy; Quality of Life; Symptom Management
MeSH Terms: conditions — Prostatic Neoplasms | interventions — saw palmetto extract

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Phase 1: The dose finding phase (DFP) (Other): Patients received Saw Palmetto Soft Gel capsules in 320mg or 640mg or 960mg to determine the maximum therapeutic dose
  Interventions: Drug: Saw Palmetto
- Phase 2: RCT phase- Saw Palmetto (Active Comparator): Patients received the predetermine the maximum therapeutic dose of Saw Palmetto Soft Gel capsules in phase 1, which is 960mg.
  Interventions: Drug: Saw Palmetto
- Phase 2: RCT phase- Placebo (Placebo Comparator): Patients received Soybean Oil Soft Gel as the placebo treatment
  Interventions: Drug: soybean oil soft gel

INTERVENTIONS:
Drug: Saw Palmetto — 1 of 3 doses of Saw Palmetto (320, 640, 960mg/day)
  Other Names: SP
  Arms: Phase 1: The dose finding phase (DFP); Phase 2: RCT phase- Saw Palmetto
Drug: soybean oil soft gel — placebo (soybean oil soft gel)
  Other Names: Placebo
  Arms: Phase 2: RCT phase- Placebo

SUMMARY:
The aim of this study is to test whether Saw Palmetto, is useful in preventing or reducing the side effects for men undergoing radiation therapy for prostate cancer. Urinary symptoms will be recorded each week, as well as assessment of quality of life through: 1) Physical Well-Being 2) Social/Family Well-being 3) Emotional Well-Being, and 4) Functional Well-Being.

DETAILED DESCRIPTION:
Lower urinary tract symptoms (LUTS) affect from 75-80% of men undergoing radiation therapy (RT) for prostate cancer. The purpose of this study was to determine the feasibility, safety and efficacy of inexpensive, non-toxic herbal supplement, Saw Palmetto (SP), in treating these distressing symptoms.

The study consisted of two phases: Dose Finding phase (DFP), and Exploratory Randomized Controlled Trail (RCT) phase. In the 12 week DFP, participants were given one of three doses (SP 320 mg, SP 640mg, and SP 960 mg) using the Time-to-Event Continual Reassessment Method to determine the maximum therapeutic dose (MTD). Once the MTD was determined the RCT phase was begun, participants were allocated to receive either the predetermined MTD (960 mg) in the DFP or a placebo to obtain preliminary evidence of efficacy of SP on LUTS.

Safety data consisted of the Common Terminology for Adverse Events criteria for nausea, gastritis, and anorexia. Efficacy of the MTD was evaluated by weekly symptom data and voiding diary. A pill diary was used to ensure the intervention fidelity.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years or older
* Adenocarcinoma of the prostate
* Serum Prostate Specific Antigent (PSA) ≤ 40ng/ml
* Combined Gleason Score ≤ 8
* Karnofsky level of performance of > 70%
* Consented to undergo definitive Radiation Therapy

Exclusion Criteria:

* Stage T4 or M1
* Patient using own supply of Saw Palmetto or any other supplement containing the following herbs: Pygeum (African Plum), Urtica Dioica (Stinging nettle), Cucurbita peponis (pumpkin seed), PC-SPES (combination of 8 herbs), Beta-sitsterol (plant sterols) or Cernilton (rye grass pollen).
* Prior pelvic radiation therapy
* Abnormality in liver and kidney function as evidenced by greater than twice the normal values of Blood Urea Nitrogen (BUN), serum creatine, serum transaminases, and alkaline phosphatase.
* Uncontrolled hypertension despite use of antihypertensive medication
* Presence of major psychiatric or medical illness (e.g., major cardiovascular events within the previous 12 months)

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gwen Wyatt, PhD, RN, Principal Investigator — MichiganState University
Locations (6):
- United States (6):
  - Allegiance Health, Jackson, Michigan
  - McLaren Greater Lansing, Lansing, Michigan
  - Sparrow Cancer Center, Lansing, Michigan
  - McLaren Macomb, Mount Clemens, Michigan
  - McLaren Central Michigan, Mount Pleasant, Michigan
  - St. Joseph Mercy Oakland Hospital, Pontiac, Michigan

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1: Saw Palmetto Soft Gel 320mg/Day: Participants in this arm received 320mg/day of Saw Palmetto Soft Gel capsules.
- Phase 1: Saw Palmentto Soft Gel 640mg/Day: Participants in this arm received 640mg/day of Saw Palmetto Soft Gel capsules.
- Phase 1: Saw Palmetto Soft Gel 960mg/Day: Participants in this arm received 960mg/day of Saw Palmetto Soft Gel capsules.
Period: Overall Study
Arm/Group | Phase 1: Saw Palmetto Soft Gel 320mg/Day | Phase 1: Saw Palmentto Soft Gel 640mg/Day | Phase 1: Saw Palmetto Soft Gel 960mg/Day | Phase 2: RCT Phase- Saw Palmetto | Phase 2: RCT Phase- Placebo
Started | 3 | 4 | 20 | 10 | 11
Completed | 3 | 3 | 16 | 6 | 9
Not Completed | 0 | 1 | 4 | 4 | 2
Not completed — Lost to Follow-up | 0 | 0 | 2 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 2 | 1
Not completed — Other | 0 | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 1: Saw Palmetto Soft Gel 640mg/Day: Participants in this arm received 640mg/day of Saw Palmetto Soft Gel capsules.
- Active Comparator: Phase 2: RCT Phase- Saw Palmetto: Patients received the predetermine the maximum therapeutic dose of Saw Palmetto Soft Gel capsules in phase 1, which is 960mg
- Placebo Comparator: Phase 2: RCT Phase- Placebo: Patients received Soybean Oil Soft Gel as the placebo treatment
- Total: Total of all reporting groups
Arm/Group | Phase 1: Saw Palmetto Soft Gel 320mg/Day | Phase 1: Saw Palmetto Soft Gel 640mg/Day | Phase 1: Saw Palmetto Soft Gel 960mg/Day | Active Comparator: Phase 2: RCT Phase- Saw Palmetto | Placebo Comparator: Phase 2: RCT Phase- Placebo | Total
Number analyzed (Participants) | 3 | 4 | 20 | 10 | 11 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (3.0) | 62.75 (12.09) | 62.1 (5.3) | 66.70 (11.30) | 67.82 (7.22) | 67.29 (9.16)
Sex/Gender, Customized [Number; unit: participants]
  Male | 3 | 4 | 20 | 10 | 11 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 3 | 4 | 14 | 8 | 8 | 37
  Unknown or Not Reported | 0 | 0 | 5 | 2 | 3 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 1 | 0 | 3
  White | 3 | 4 | 15 | 9 | 10 | 41
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 3 | 0 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 20 | 10 | 11 | 48

OUTCOME MEASURES:

1. Primary Outcome: Feasibility
Description: Assess a Saw Palmetto supplementation protocol for feasibility by evaluation if at least 70% of eligible men consent, and if at least 70% of men enrolled at each dose complete the study.
Time Frame: Baseline to Week 12 for each phase.
Population: Number of men who started
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1: Men in 320mg/Day DFP: Men assigned to the 320mg/Day group in the dose finding phase.
- Phase 1: Men in 640mg/Day DFP: Men assigned to the 640mg/Day group in the dose finding phase.
- Phase 1: Men in 960mg/Day DFP: Men assigned to the 960mg/Day group in the dose finding phase.
- Phase 2: Saw Palmetto 960 mg RCT: Men assigned to the 960mg/Day of Saw Palmetto in the pilot RCT Phase
- Phase 2: Placebo RCT: Men assigned to the placebo in the pilot RCT Phase
Arm/Group | Phase 1: Men in 320mg/Day DFP | Phase 1: Men in 640mg/Day DFP | Phase 1: Men in 960mg/Day DFP | Phase 2: Saw Palmetto 960 mg RCT | Phase 2: Placebo RCT
Number analyzed (Participants) | 3 | 4 | 20 | 10 | 11
Participants | 3 | 3 | 16 | 6 | 9

2. Primary Outcome: Efficacy
Description: Evaluate preliminary efficacy of Saw Palmetto at the MTD as compared to the placebo group with respect to Health-Related Quality of life (HRQOL) including physical functioning and symptoms. The outcomes were measured using 1) the International Prostate Symptoms Score (IPSS) and 2) the total and subscales of the Functional Assessment of Cancer Therapy-Prostate (FACT-P). The IPSS which ranges from 0-35. A lower score indicates better symptoms. The FACT-P has the following subscores and ranges: emotional well-being (0-24), functional well-being (0-28), physical well-being (0-28), social well-being (0-28), and prostate-specific concerns (0-48). The FACT-P total is comprised of the sum of the subscales and ranges from 0-156. For the FACT-P, a higher score indicates better quality of life. Each values was created as an average over time from a linear mixed effects model that adjusted for baseline values.
Time Frame: HRQOL: Baseline, week 12, 14, & 22. IPSS: Baseline, week 3-12, 14, & 22.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phase 2: RCT Phase- Saw Palmetto | Phase 2: RCT Phase- Placebo
Number analyzed (Participants) | 6 | 9
units on a scale
  IPSS | 10.54 (1.29) | 9.41 (1.21)
  FACT-P total | 124.77 (4.37) | 124.48 (4.18)
  FACT-P emotional well-being | 20.77 (0.84) | 21.62 (0.79)
  FACT-P functional well-being | 22.24 (1.30) | 21.20 (1.25)
  FACT-P physical well-being | 24.00 (0.86) | 25.67 (0.81)
  FACT-P social well-being | 23.38 (1.08) | 21.02 (1.01)
  FACT-P Prostate specific concern | 35.13 (1.92) | 33.81 (1.82)

3. Primary Outcome: Number of Participants With Dose Limiting Toxicities to Determine the Maximum Tolerated Dose
Description: Dose limiting toxicities was defined as the Common Terminology Criteria for Adverse Events (CTCAE) Grade 2 or higher for gastrointestinal symptoms (nausea, gastritis, anorexia). The maximum tolerated dose (MTD) was established among 320mg, 640mg,or 960mg, at which less than 10% of men report less than a grade 2 of gastrointestinal symptoms.
Time Frame: Baseline to Week 12
Population: Number of participants reporting adverse events at grade 2 or higher, according to the TITE-CRM algorithm
Measure: Number; unit: participants
Groups:
- Phase I: Saw Palmetto Soft Gel 640mg/Day: Participants in this arm received 640mg/day of Saw Palmetto Soft Gel capsules.
- Phase I: Saw Palmetto Soft Gel 960mg/Day: Participants in this arm received 960 mg/day of Saw Palmetto Soft Gel capsules.
Arm/Group | Phase 1: Saw Palmetto Soft Gel 320mg/Day | Phase I: Saw Palmetto Soft Gel 640mg/Day | Phase I: Saw Palmetto Soft Gel 960mg/Day
Number analyzed (Participants) | 3 | 3 | 16
participants | 0 | 0 | 0
Statistical Analysis 1: Comparison: Phase 1: Saw Palmetto Soft Gel 320mg/Day vs Phase I: Saw Palmetto Soft Gel 640mg/Day vs Phase I: Saw Palmetto Soft Gel 960mg/Day; The time-to-event continual reassessment method (TITE-CRM) was used The TITE-CRM incorporated a decision rule for the allocation of next participant to a dose of SP based on the current estimate of toxicity. The first men were allocated to lowest dose (320 mg); when no adverse event was reported during 12 weeks, the dose was increased to 640 mg for next men, and then to 960 mg in the absence of advert event; Test type: Other; Maximum Tolerated Dose (MTD) = 960

ADVERSE EVENTS:
Time Frame: Adverse events were tracked with the Common Terminology Criteria for Adverse Events (CTCAE) at weeks 1 (baseline), 2-12, 14, 22 and 62.
Description: Adverse events were tracked with the Common Terminology Criteria for Adverse Events (CTCAE) including anorexia, nausea, gastritis, hematuria, hemorrhoids, diarrhea, proctitis, pruritis/itching, and fatigue.
Groups:
- Phase 2: RCT Phase- Saw Palmetto: Patients received the predetermine the maximum therapeutic dose of Saw Palmetto Soft Gel capsules in phase 1, which is 960 mg.
Arm/Group | Phase 1: The Dose Finding Phase (DFP) | Phase 2: RCT Phase- Saw Palmetto | Phase 2: RCT Phase- Placebo
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 0/27 | 0/10 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No